CLINICAL TRIAL: NCT04662775
Title: Formative Evaluation of a Home-based Physical Activity Intervention for Adolescent Girls - The HERizon Project: A Randomised Controlled Trial
Brief Title: Formative Evaluation of The HERizon Project
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Liverpool John Moores University (Other)
Collaborators: University of Liverpool (Other); Dublin City University (Other); Radboud University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HERizonProject
Record Dates: First submitted 2020-11-27; First posted 2020-12-10 (Actual); Last update posted 2020-12-16 (Actual); Status verified 2020-11

CONDITIONS: Physical Activity
Keywords: physical activity; adolescents; girls; behaviour change; qualitative
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Intervention Model Description: Block randomisation with country-level stratification was used using Microsoft Excel to allocate the participants on entry (1:1 ratio to groups)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): This group received the multi-component physical activity intervention (physical activity programme, weekly behaviour change support calls, non-reply text messages)
  Interventions: Behavioral: HERizon Project
- Waitlist control (No Intervention): Participants in the wait-list control group were asked to continue their usual PA habits and received no additional contact from the research team outside of data collection points. Following post-intervention data collection, control group participants were invited to participate in the same intervention as described above.

INTERVENTIONS:
Behavioral: HERizon Project — 1. Participants were asked to complete 3x30-minute physical activity sessions each week & record their sessions using a logbook. They were given the choice of different types of home-based virtual exercise. 2. Behaviour change support calls - participants were allocated an "Activity Mentor" (trainee sport and exercise psychologists, was supervised by a HCPC-registered Psychologist). Participants had seven weekly videocalls. Each call was based on a pre-planned session outline and was goal orientated, participant centred and focused on physical activity. 3. No reply SMS - Participants received 3 standardised text messages each week, aimed at providing physical activity -related facts, encouragement and study information.
  Arms: Intervention group

SUMMARY:
This mixed methods study was the feasibility phase of a broader intervention of research (The HERizon Project) that aims to develop a theory-based physical activity intervention targeting adolescent girls in the UK and Ireland. The design was a two-arm randomised controlled trial, comprising of (i) the HERizon six week remote intervention arm and (ii) a wait-list control arm. Block randomisation with country-level stratification was used to allocate the participants on entry. The primary outcome of the study was change in moderate to vigorous physical activity levels. Secondary outcomes included cardiorespiratory fitness, muscular strength and endurance, exercise motivation, perceived competence, self-esteem and body appreciation. Assessments were conducted pre-intervention (April/May, 2020) and repeated immediately post-intervention (June/July, 2020). As the study ran during the COVID-19 pandemic, all participants began the intervention in full national lockdowns, with all local schools and amenities being closed. Restriction began to be lifted in the last week of June in Ireland and in the first week of July in the UK, with some local amenities opening and small outside group gathering being permitted. Due to the nature of the study, participants and project deliverers could not be blinded to the assigned intervention.

DETAILED DESCRIPTION:
Design. This physical activity study will be evaluated using a two-arm randomised controlled trial with an intervention group and a wait-list control group. Assessments will be conducted at baseline and 6 weeks from baseline. Assessments will occur remotely in the participants' homes in April/May (baseline) and May/June (end point).

Recruitment. We aim to recruit 40 participants by convenience sampling through links with secondary school teachers, LJMU communications with staff and students, and via social media. The participant information sheet will be emailed to all potential participants. The email will ask potential participants to read the attached information sheet and they will be encouraged to ask the researchers questions. Participants will have up to one week to decide if they would like to participate in the study. Online consent forms will be used to obtain written informed consent for both the participant and their parent/ guardian. Participants will be given a link where they can sign the document online or they can sign a paper form and scan a copy back to the researcher. Participants will also be asked to provide verbal consent before any phone interviews and to tick a box confirming their consent before completing any questionnaires.

Randomisation. Using a computer-based randomisation tool, participants will be assigned to one of the two arms (intervention or wait list control). To make allocation more time efficient, randomisation will occur prior to baseline assessment. Once the follow up assessment has taken place for the intervention group, the wait-list control participants can begin the six-week physical activity programme.

Intervention. Due to the current COVID-19 pandemic, all aspects of this research project will be conducted virtually and adhere to the UK Government advice at the time the intervention begins. Assessments will be carried out as self-assessments by the participants in both the wait-list control and the intervention group in their own homes at two time points (week 0 and 6). The goals of this physical activity programme are to 1) inform participants of specific behaviours change skills related to adopting and maintaining a physically active life during and after the COVID-19 pandemic (e.g. self-monitoring, goal setting and overcoming challenges), and 2) increase adolescent girls' habitual physical activity (steps per day). To achieve these goals the following elements will be implemented:

* Exercise Sessions: Participants will be given the choice of different types of home-based virtual exercise videos, e.g. boxercise, dance classes, Pilates, bodyweight resistance exercise, Joe Wicks Body Coach YouTube channel, or design their own using a home-based exercise booklet with a choice of body weight exercises (booklet attached in appendix). Participants will be asked to complete 3 sessions of 30 minutes per week. The researcher will host an online group fitness class each week which participants are also invited to join. This option is to allow participants to engage in the social elements of physical activity but from the comfort of their own homes. It is also thought that having a scheduled set time to join a class may increase motivation and improve adherence, however this is optional. Participants will have the flexibility to choose whatever type of exercise suits their preferences and abilities. Using a printed or online template (participant preference), participants are asked to record what activity they did, the duration and a reflection of how they found the workout e.g. more motivated in the morning, burpees really difficult, enjoy a mix of aerobic and resistance training.
* Behaviour Change Calls: Weekly by phone call or video conference (at the preference of the participant e.g. Skype or Zoom) by a trained Prof Doc psychology candidate. Behaviour change support is based on self-determination principles (autonomy, competence and relatedness). Each call will be based on a pre-planned session outline and will be goal orientated, participant centred and focused on PA. Calls are expected to last 15-20 minutes per participant.
* No Reply SMS: Sent to the participant's mobile phone twice per week by a trained Prof Doc psychology candidate from an online messaging software (this option will be used as given the current situation researchers cannot access LJMU phones. This service is password protected and participants phone numbers will not be stored online). All messages will be standardised (not personally tailored) and will be focused on behaviour change techniques or reminders.

Control: Participants in the wait-list control group will receive the physical activity programme after follow-up measures have been taken from the intervention group. Participants in the control group will only have contact with the research team during data collections for the first six week (and then will carry out six weeks with prof doc behaviour change support and SMS support). They will then complete all self-assessment measures at week 0 and 6 (self-report and objective physical activity levels, aerobic capacity, muscular endurance, strength/power, PA motivation, self-esteem, body appreciation and PA competence).

Primary and Secondary Outcomes The assessment of the primary and secondary outcomes will be conducted without on-site presence of the participants or researchers at two occasions; baseline (week 0) and post-intervention (week 6). Self-reported and objectively assessed PA levels of one week , and psychosocial determinants of physical activity will be assessed at baseline and post-intervention (week 0 and week 6). At 6 weeks, a sub-group of participants will be asked to do phone interviews with the lead researcher to give their feedback on the intervention.

Phone interviews. Interviews will be conducted with a random subsample of 10 participants from the intervention group at week 6. Interviews will be conducted via phone call and will last approximately 20-30 minutes. Discussion will focus on participants' experience of the intervention, suggestions, perceived benefits of the intervention and perceived facilitators and barriers (i.e. what worked well, what worked less well). Qualitative measures are vital to this study as is it important to collect adolescents' perspectives of data collection measures, the method of behaviour change support and the virtual exercise. Through interviews we hope to gain a rich insight into their perceived barriers and facilitators to the PA programme. By gaining this invaluable knowledge the programme can be further refined for future implementation. Considerations have been outlined in regard to what the researcher might do in the unlikely event of a child disclosing potentially concerning information.

Procedures. Written informed consent from participants and parents/guardians will be returned to the researcher prior to the commencement of testing. Testing will occur in the participants home remotely. It is advised that participants complete the testing, exercise sessions and behaviour change support calls in a public area of their home but in private e.g. in the sitting room and are not permitted to take any calls from the research team or prof doc candidates in their bedrooms. Following written consent, participants will complete all questionnaires online (approximately 30 minutes) - self-reported physical activity, sociodemographic and psychosocial determinants. Participants will then complete the fitness measures using the RTFT app (30 minutes). Participants will monitor their steps using a mobile-based app for 7 days before starting their 6-week physical activity programme. In total assessments should take approximately one hour and will be conducted at baseline (week 0) and post-intervention (week 6).

Each week for six weeks, participants will; (1) complete three 30-minute exercise sessions, (2) receive two behaviour change support SMS to their mobile from an LJMU prof doc for six weeks, e.g. motivation or reminder texts, (3) have one 15-20-minute call with an LJMU prof doc each week for six weeks. This will be done via phone call or video call (at the participants' preference) and will focus on behaviour change support, e.g. goal setting and overcoming challenges. The exercise options the girls can choose from are based on the results of previously conducted focus groups with a different cohort of adolescent girls from the UK and Ireland, i.e. their favourite types of activity were home-based, video-led, boxing, dancing and a mix of aerobic and resistance exercises. Participants adherence will be monitored in two ways, a. written self-reported exercise log and b. during weekly support call with prof doc.

Data Processing and Statistical Analyses. Participants' baseline characteristics will be presented as means (standard deviation) for all continuous variables and as percentages for categorical variables. Statistical tests, including t-tests, Mann-Whitney tests and Pearson's chi-squared or Fisher's exact test will be used, as appropriate, to investigate any differences in demographic factors between the two groups. Linear missed models will be used to compare groups, time and group x time interaction. Recruitment and retention will also be summarised descriptively. Multilevel modelling will be used to assess preliminary effectiveness of the intervention on adolescents PA. Statistical analysis of measured outcomes will be conducted using the latest edition of SPSS Statistics (SPSS Inc., IBM Corp., Armonk, NY).

All semi-structured interviews will be audio recorded and transcribed verbatim by the primary researcher (when they will then be anonymised). Thematic analysis will be conducted using NVivo electronic software to identify common themes and sub-themes (Braun & Clarke, 2002).

ELIGIBILITY:
Inclusion Criteria:

* Female
* 13-16 years
* Living in the UK and Ireland
* Ability to participate in moderate intensity physical activity according to the Physical Activity Readiness Questionnaire

Exclusion Criteria:

* Currently pregnant
* Severe psychological or neurological condition
* No access to a phone or computer

Ages: 13 Years to 16 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 42 (Actual)
Dates: Start 2020-04-15 (Actual); Primary Completion 2020-07-08 (Actual); Study Completion 2020-07-08 (Actual)

PRIMARY OUTCOMES:
Physical activity | 6 weeks
  Moderate to vigorous physical activity was assessed using the 8-item sub-scale World Health Organisation Health Behaviours of School Children questionnaire which has been validated with adolescents. This was used to collect self-reported physical activity over the previous seven-day period at baseline and post-intervention. Girls self-reported the estimated hours they spent engaging in physical activity before school, during school, after school and at weekends. The total hours spent in moderate to vigorous physical activity were then averaged across the week to find daily averages. The government guidelines are 60 minutes per day of physical activity on average across the week.

SECONDARY OUTCOMES:
Cardiorespiratory fitness | 6 weeks
  The 20-metre progressive shuttle run test (20mSRT) was used to provide an estimate of cardiorespiratory fitness. Participants ran back and forth between two markers positioned 20 meters apart at a pace signalled by an audio file on the Resistance Training for Teens (RTT) app. The test starts at a pace of 8.5 kmph and gradually increases in 0.5 kmph increments as the levels progress (pace increases approximately every minute). The test ended when the participant could not make it to a line for two consecutive beeps and the final successful stage was recorded using the app. Parents were instructed to provide verbal encouragement throughout the test with the aim of girls reaching volatile exhaustion. This test has been validated with adolescents previously.
Muscular endurance | 6 weeks
  A 90-degree push up test was used as a measure of upper body muscular endurance. Using an audio file on the RTT app, participants performed push ups at a cadence of 40 bpm. Participants began in a high plank position (hands positioned under the shoulders, toes touching the floor, back in a straight line) and lowered themselves to the ground in a controlled manner until their arms are at a 90-degree angle from which they then pushed back up and returned to a high plank position. Parents counted and recorded the number of push ups and the test was terminated if participants could not maintain correct exercise form or voluntarily stopped. The push up test has been validated as a measure of muscular endurance with adolescents.
Muscular strength | 6 weeks
  A standing long jump test was used as a measure of lower body muscular strength. Participants began standing with their toes behind a starting marker and then performed a long jump, jumping from and landing on two feet. A parent/ guardian recorded the distance travelled from starting marker to the participant's foot in the landing position. Participants completed this measure twice with the longest jump being recorded as the final score. The long jump test has been found to be a valid and reliable measure of adolescents' muscular strength.
Exercise motivation | 6 weeks
  The Behavioural Regulation in Exercise Questionnaire 3 (BREQ-3) combines 19-items from the BREQ-2 , four additional integrated regulation items (validated by Wilson et al., 2006]), and one additional introjected regulation item. The questionnaire contains six subscales, ranging from amotivation, through controlled motivation (external regulation, introjected regulation) to autonomous motivation (identified regulation, integrated regulation, intrinsic motivation). Participants were scored using a five-point Likert scale ranging from "Not true (0)" to "True (4)". Higher scores indicate a higher motivation within that specific sub-scale.
Body image | 6 weeks
  Body image was measured by the 10-item Body Appreciation Scale which was also scored using a five-point Likert scale ranging from "Never (0)" to "Always (4)". Questions include statements such as "I respect my body" and "I feel love for my body". Higher scores reflect a higher level of body appreciation. Responses demonstrated excellent internal consistency (Cronbach's alpha between 0.94 to 0.95).
Competence | 6 weeks
  PA competence was measured by an adapted 4-item Perceived Competence Scale which was scored using a seven-point Likert scale ranging from "Strongly disagree (1)" to "Strongly agree (7)". Questions include "I am capable of being physically active regularly". Higher scores indicate a higher perceived competence in PA. Responses within our sample demonstrated excellent internal consistency (Cronbach's alpha between 0.85 to 0.91).
Self-esteem | 6 weeks
  Self-esteem was measured by the 12-item Adolescent Self-Esteem Questionnaire which was scored using a five-point Likert scale ranging from "Almost all of the time (1)" to "Hardly ever (5)". Questions include "I feel I can be myself around other people". A higher score indicates a higher level of self-esteem. To generate an overall score for each questionnaire, questions were scored using the corresponding Likert scale and a mean score was then calculated. Responses within our sample demonstrated acceptable internal consistency (Cronbach's alpha between 0.68 to 0.72).
Daily step count | 6 weeks
  A mobile phone based pedometer app (Google Fit) was used to record participants' steps for seven-days at baseline and post-intervention. Steps for the seven-days were averaged to calculate a mean daily step score. Girls were instructed to keep their mobile phone on their person as much as possible over the seven-day period, e.g. in their pocket. Mobile pedometers have been validated in adolescents.
Sedentary behaviour | 6 weeks
  Sedentary behaviour was assessed using the 8-item sub-scale World Health Organisation Health Behaviours of School Children questionnaire which has been validated with adolescents. Participants estimated the minutes spent in sedentary behaviour whilst watching television, playing video games or using the internet. This was used to collect self-reported physical activity over the previous seven-day period at baseline and post-intervention. The total minutes spent in sedentary behaviour were then averaged across the week to find daily averages. Sedentary time should be limited to a maximum of two hours per day.

CONTACTS AND LOCATIONS:
Overall Officials: Anton Wagenmakers, Principal Investigator — Liverpool John Moores University
Locations (3):
- Dublin City University, Dublin, Ireland
- United Kingdom (2):
  - LiverpoolJMU, Liverpool, Merseyside
  - Wolfson Centre for Personalised Medicine, Institute of Systems, Molecular and Integrative Biology, Liverpool

IPD SHARING:
Plan to Share IPD: No
Participant data will only be accessible to the research team and will be destroyed after 5 years as per university policy. All personal data will be anonymised using a participant code. Should a participant want access to their data will may ask for a copy at any time point.